CLINICAL TRIAL: NCT02476695
Title: Research on FibroTouch Noninvasive Evaluation of Liver Fibrosis and Cirrhosis
Brief Title: FibroTouch Non-invasive Evaluation of Liver Fibrosis and Cirrhosis
Status: Completed | Type: Observational
Sponsor: Wuxi Hisky Medical Technology Co Ltd (Industry)
Collaborators: Beijing Friendship Hospital (Other); The Military General Hospital of Beijing, PLA (Unknown); The First Affiliated Hospital, Third Military University (Unknown); The First Affiliated Hospital of the Fourth Military Medical University (Other); The First Hospital of Jilin University (Other); Hebei Medical University Third Hospital (Other); Henan Provincial People's Hospital (Other); Jiangsu Provincial People's Hospital (Other); Ruijin Hospital (Other); West China Hospital (Other); Tianjin Third Central Hospital (Other); No.85 Hospital, Changning, Shanghai, China (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other); Hospital of Chinese Medicine of the Xinjiang Uygur Autonomous Region (Unknown); The China-Japan Friendship Hospital (Unknown); Peking University Clinical Research Institute (PUCRI) (Unknown)
Responsible Party: Sponsor
Other Study IDs: ChiCTR-DDT-14004429
Record Dates: First submitted 2015-05-25; First posted 2015-06-19 (Estimated); Results first posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Liver Fibrosis; Cirrhosis; Chronic Hepatitis B
Keywords: CHB
MeSH Terms: conditions — Liver Cirrhosis; Fibrosis; Hepatitis B, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (4):
- S0/1: S0 = no fibrosis and S1 = portal fibrosis without septa
  Interventions: Device: FibroTouch Examination; Device: FibroScan Examination; Device: Ultrasonic B Examination
- S2: S2 = portal fibrosis with few septa
  Interventions: Device: FibroTouch Examination; Device: FibroScan Examination; Device: Ultrasonic B Examination
- S3: S3 = numerous septa without cirrhosis
  Interventions: Device: FibroTouch Examination; Device: FibroScan Examination; Device: Ultrasonic B Examination
- S4: S4 = liver cirrhosis (compensatory stage)
  Interventions: Device: FibroTouch Examination; Device: FibroScan Examination; Device: Ultrasonic B Examination

INTERVENTIONS:
Device: FibroTouch Examination — Liver stiffness measurements are performed using FibroTouch and the procedure is non-invasive and painless.
Device: FibroScan Examination — Liver stiffness measurements are performed using another transient elastography, FibroScan, and the procedure is non-invasive and painless.
Device: Ultrasonic B Examination — The ultrasonic B examination is made at an empty stomach for ≥8h. The inner diameter of liver, spleen, gallbladder, portal vein and splenoportal vein is measured through the ordinary two-dimensional ultrasonic examination. The echo data of liver surface/edge/parenchyma and gallbladder wall is scored to evaluate the severity of fibrosis.

SUMMARY:
This prospective and multicenter study is to determine the diagnostic performance (accuracy, specificity and sensitivity) of transient elastography (FibroTouch) for liver fibrosis assessment in chronic hepatitis B (CHB) patients using ROC analysis, and liver biopsy as the reference.

Actual 517 patients will be enrolled to guarantee 500 final statistical cases; and ≥100 cases are required for fibrosis stage S0/1, S2, S3 and S4 (compensatory stage of cirrhosis), respectively. For each stage, the case is assigned as equally as possible.

DETAILED DESCRIPTION:
The liver diseases frequently occur in China. For various reasons, the chronic liver diseases are not controlled in time, and then develop gradually into liver fibrosis and cirrhosis. Without effective treatment, the advanced liver cirrhosis seriously influences the quality of patients' life, and places an intolerable burden on family and society. At present, the scholars generally thought that the liver fibrosis at early stages is reversible. Therefore, if the liver fibrosis in patients with chronic liver diseases can be accurately evaluated at early stages and be treated in time, so we can stop the progress of diseases and reduce the occurrence of liver cirrhosis and liver cancer.

For many years, liver biopsy is still as "golden standard" for diagnosis of liver inflammation and fibrosis. However, with its invasiveness, potential risks and some complications, liver biopsy is limited in clinical application due to the poor acceptability and repeatability. In recent years, the liver fibrosis cannot directly and accurately diagnose via the various diagnostic models using serological biomarkers (e.g. FIBROTEST and APRI) and medical imaging technologies (e.g. ultrasonic B, CT and MRI).

Transient elastography is a new technology in the field of ultrasonic imaging. Liver stiffness measurement (LSM) is based on the relationship between the speed of spread of acoustic wave in tissues and stiffness of the tissues. It utilizes specific probes to send out controlled low-frequency shear waves, the waves signals transmit through liver tissues, a high-frequency signals will track the transmitting process of shear wave in the liver and the value of liver stiffness (kPa) is quickly calculated with reference to a built-in liver histological model, which provides a quantitative standard for diagnosis of liver fibrosis of chronic liver disease. The bigger LSM value means the faster transmission of shear wave, and the harder of determined liver tissue.

As stated in the "12th Five-year Plan for Medical Device Technological Industry" (the Ministry of Science and Technology), China will greatly support the research and development of new medical devices and promote the application of Chinese transient elastography system, FibroTouch, which was R&D by Tsing-Hua University independently with new algorithm. FibroTouch can rapidly determine the LSM in a non-invasive way and provide useful information for liver fibrosis and steatosis staging.

Due to FibroTouch is a new transient elastography system in marketing, there is no too much studies on the correlation between FibroTouch and liver biopsy in diagnosis of liver fibrosis and cirrhosis.

The goal of this prospective and multicenter study is to determine the diagnostic performance (accuracy, specificity and sensitivity) of FibroTouch for liver fibrosis assessment in chronic hepatitis B (CHB) patients using ROC analysis, and liver biopsy as the reference.

Actual 517 patients will be enrolled to guarantee 500 final statistical cases; and ≥100 cases are required for fibrosis stage S0/1, S2, S3 and S4 (compensatory stage of cirrhosis), respectively. For each stage, the case is assigned as equally as possible.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with age 18-65 years, both gender
* Subjects with history of HBV or HBsAg positive > 6 months up to enrollment
* Subjects with qualified liver biopsy specimens within three months (before or after) of Fibrotouch examination for pathological staging
* Subjects without chemical therapy history of powerful medicine to lower enzyme in the two weeks before blood biochemistry tests (e.g. dimethyl diphenyl bicarboxylate and bicyclol)
* Subjects must agree and sign the informed consent form

Exclusion Criteria:

* Subjects who are unable or unwilling to sign informed consent form
* Subjects who have merger of hepatitis C, alcohol and non-alcoholic fatty liver diseases, autoimmune liver diseases, inherited metabolic liver diseases, biliary systemic diseases or liver and gall parasitic diseases
* Subjects who have other serious chronic disorders or history of malignancy
* Subjects with ALT ≥5 ULN in the past 1 month
* Subjects with WBC<3.5×10^9/L, PLT<60×10^9/L, PTA<60%
* Subjects with DBIL≥1.5 ULN
* Subjects with decompensated cirrhosis (especially the people with ascites)
* Pregnant or lactating women, or women who has a pregnant plan and don't want to birth control in the study period
* Subjects who have wound on the right upper abdomen recently
* Subjects who have various space-occupying tumor or cyst in right liver
* Subjects who have none or limited legal capacity

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subjects with chronic hepatitis B (CHB), who underwent a liver biopsy in hospital and meets all of the inclusion criteria and none of the exclusion criteria, may participate in this study. Within three months of FibroTouch examination, subjects are required to have qualified histological specimens of liver biopsy for analysis and comparison.
Sampling Method: Non-Probability Sample
Enrollment: 412 (Actual)
Dates: Start 2014-05; Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jidong JIA, MD, Study Chair — Beijing Friendship Hospital; Jianbiao CAO, MD, Principal Investigator — The Military General Hospital of Beijing, PLA; Qing MAO, MD, Principal Investigator — The First Affiliated Hospital, Third Military University; Ying HAN, MD, Principal Investigator — The First Affiliated Hospital of the Fourth Military Medical University; Junqi NIU, MD, Principal Investigator — The First Hospital of Jilin University; Yuemin NAN, MD, Principal Investigator — Hebei Medical University Third Hospital; JIA SHANG, MD, Principal Investigator — Henan Provincial People's Hospital; Jun LI, MD, Principal Investigator — Jiangsu Provincial People's Hospital; Qing XIE, MD, Principal Investigator — Ruijin Hospital; Hong TANG, MD, Principal Investigator — West China Hospital; Tao HAN, MD, Principal Investigator — Tianjin Third Central Hospital; Qingchun FU, MD, Principal Investigator — No.85 Hospital, Changning, Shanghai, China; Zhiliang GAO, MD, Principal Investigator — Third Affiliated Hospital, Sun Yat-Sen University; Xiaozhong WANG, MD, Principal Investigator — Hospital of Chinese Medicine of the Xinjiang Uygur Autonomous Region; Anlin MA, MD, Principal Investigator — The China-Japan Friendship Hospital
Locations (15):
- China (15):
  - Beijing Friendship Hospital, Capital Medical University, Beijing
  - The China-Japan Friendship Hospital, Beijing
  - The Military General Hospital of Beijing, PLA, Beijing
  - The First Bethune Hospital of Jilin University, Changchun
  - West China Hospital, Sichuan University, Chengdu
  - The First Affiliated Hospital, Third Military University, Chongqing
  - The Third Affiliated Hospital of Sun Yat-Sen University, Guangzhou
  - Jiangsu Provincial People's Hospital, Nanjing
  - No.85 Hospital of the PLA, Shanghai
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai
  - The Third Hospital, Hebei Medical University, Shijiazhuang
  - Tianjin Third Central Hospital, Tianjin
  - Hospital of Chinese Medicine of the Xinjiang Uygur Autonomous Region, Ürümqi
  - The First Affiliated Hospital, Fourth Military University, Xi'an
  - Henan Provincial People's Hospital, Zhengzhou

RESULTS

PARTICIPANT FLOW:
Groups:
- All Enrollment Patients: Patients with chronic hepatitis B who underwent a liver biopsy and LSMwere considered for enrollment.
  F0, no fibrosis; F1, portal fibrosis without septa; F2, portal fibrosis and a few septa; F3, numerous septa without cirrhosis; and F4, cirrhosis.
  Clinical and laboratory investigations; Non-invasive serum markers of liver fibrosis; LSM by FibroTouch transient elastography; Assessment of liver pathology
Period: Overall Study
Arm/Group | All Enrollment Patients
Started | 412
F0 | 11
F1 | 162
F2 | 118
F3 | 95
F4 | 26
Completed | 412
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Patients With Chronic Hepatitis B: The METAVIR scoring system classifies liver fibrosis in five stages as follows: F0=no fibrosis F1 = portal fibrosis without septa F2 = portal fibrosis with few septa F3 = numerous septa without cirrhosis F4 = liver cirrhosis (compensatory stage)
  Clinical and laboratory investigations; Non-invasive serum markers of liver fibrosis; Non-invasive serum markers of liver fibrosis; Assessment of liver pathology
Arm/Group | Patients With Chronic Hepatitis B
Number analyzed (Participants) | 412
Age, Continuous [Mean (Standard Deviation); unit: years] — Measure Analysis Population Description: 412 participants were analysed in total, not in different groups.
  years | 39.4 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 276
  Male | 136
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 412
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: The Clinical Value Evaluation of FibroTouch for Non-invasive Diagnosis of Liver Fibrosis in Patients With Chronic Hepatitis B by Using Liver Pathology as the Gold Standard for Judging CHB Liver Fibrosis Stage
Description: Altogether 412 patients were included to analyze the diagnostic performance of FibroTouch. The area under the receiver operating characteristic curve for the LSM was 0.846 (95% confidence interval CI 0.808-0.880) for fibrosis stage ≥ F1, 0.850 for ≥ F2, 0.908 for ≥ F3 and 0.874 for F4. Optimal LSM cut-off values for diagnosing fibrosis stage ≥ F1, ≥ F2, ≥ F3, and F4 were 5.5 kPa, 7.85 kPa, 10.0 kPa, and 12.7 kPa, respectively.
Time Frame: Participants will be offered a FibroTouch examination before or after taking the test of liver biopsy, and the time interval should not exceed 3 months.
Population: ROC analysis is based on a binary classification model, which refers to models with only two types of output results, such as: (positive/negative) (diseased/not diseased).Due to the particularity of this analysis method, there is no ROC value for F0.
Measure: Number (95% Confidence Interval); unit: probability
Groups:
- F1 Fibrosis Stage: Patients in F1 fibrosis stage，by liver biopsy
- F2 Fibrosis Stage: Patients in F2 fibrosis stage，by liver biopsy
- F3 Fibrosis Stage: Patients in F3 fibrosis stage，by liver biopsy
- F4 Fibrosis Stage: Patients in F4 fibrosis stage，by liver biopsy
Arm/Group | F1 Fibrosis Stage | F2 Fibrosis Stage | F3 Fibrosis Stage | F4 Fibrosis Stage
Number analyzed (Participants) | 162 | 118 | 95 | 26
probability | 0.846 [0.808 to 0.880] | 0.850 [0.811 to 0.883] | 0.908 [0.876 to 0.934] | 0.874 [0.836 to 0.903]

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Patients in F0 Fibrosis Stage: fibrosis stage：F0, by liver biopsy
- Patients in F1 Fibrosis Stage: fibrosis stage：F1, by liver biopsy
- Patients in F2 Fibrosis Stage: fibrosis stage：F2, by liver biopsy
- Patients in F3 Fibrosis Stage: fibrosis stage：F3, by liver biopsy
- Patients in F4 Fibrosis Stage: fibrosis stage：F4, by liver biopsy
Arm/Group | Patients in F0 Fibrosis Stage | Patients in F1 Fibrosis Stage | Patients in F2 Fibrosis Stage | Patients in F3 Fibrosis Stage | Patients in F4 Fibrosis Stage
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/162 | 0/118 | 0/95 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/162 | 0/118 | 0/95 | 0/26
Other Adverse Events (participants affected / at risk) | 0/11 | 0/162 | 0/118 | 0/95 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-04-17): https://cdn.clinicaltrials.gov/large-docs/95/NCT02476695/Prot_SAP_000.pdf